CLINICAL TRIAL: NCT06798766
Title: Reducing Health Inequities Through Improved Guidance and Assessment on the Early Identification of Skin Changes Associated With Chronic Venous Insufficiency (CVI) in People With Dark Skin Tones
Brief Title: Reducing Skin Tone Inequities in Chronic Venous Insufficiency
Status: Recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); University of Surrey (Other)
Responsible Party: Sponsor
Other Study IDs: EDGE reference 175656; IRAS Number 350871 (Other: Integrated research application system (IRAS))
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-01

CONDITIONS: Chronic Venous Insufficiency, CVI; Chronic Venous Insufficiency C2 or Higher; Chronic Venous Disease of Lower Limbs; Venous Leg Ulcer (VLU)
Keywords: health inequities; skin tone inequities; health equality; skin tone equality; skin assessment; physical examination; patient journey; patient experience
MeSH Terms: conditions — Blindness, Cortical; Varicose Ulcer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Work-package 1 - Mapping patient journeys and patient experiences: Participating in semi-structured interview exploring patient experience and patient journey of people with dark skin tones living with chronic venous insufficiency in the U.K.
  Number of people: 36
- Work package 2 - Informing skin assessment technique and medical photography: People with dark skin tones and known chronic venous insufficiency with up to date scan results of their blood flow seen by our trust partner (the hub of the southeast Thames vascular network) by either acute or community services.
  Number of people: 15

SUMMARY:
The aim of this project is to define assessment criteria for chronic venous insufficiency (CVI) in people with dark skin tones. It will inform future interventions and modifications to practice for the assessment of CVI in people with dark skin tones in a nurse led intervention to improve patient assessment.

To achieve this there will be two parts to this study.

1. We will explore patient journeys and patient experiences of people with dark skin tones diagnosed with chronic venous insufficiency. From this we will learn from people with dark skin tones about how they recognised skin changes in their lower legs to further inform clinical assessment guidance and techniques. We will also listen to their patient journey to identify what areas worked well and what could be developed. This will help us plan how care could be improved for similar people.
2. We will record how skin changes look and feel in people with dark skin tones and known venous disease, and photograph this. We will consider whether some additional techniques used in practice to look and feel the skin is useful and whether changing the colour balance and manipulating the photographs is useful to see these skin changes.

DETAILED DESCRIPTION:
Work-package 1 - Mapping patient journeys and patient experiences 1.1 Objective

The objective of this work package is to:

• Explore patient journeys and patient experiences of people with dark skin tones diagnosed with chronic venous insufficiency.

1.2 Purpose Patient journeys will be used as a catalyst for change in the identification of CVI for people with dark skin tones. We also aim to learn from people with dark skin tones about how they recognised skin changes in their lower legs to further inform clinical assessment guidance and techniques.

1.3 Study design This part of the study is a qualitative interview study. This design ensures patients experience from their perspectives are captured.

Mapping the clinical journey from the patient perspective has significant potential to inform the redesign of new, patient centred models of care and service delivery and understanding delays in diagnosis. The areas identified within the interviews will enable future interventions to target failures in current clinical care and the narratives of patient experiences captured within the interviews will also be recorded to form the basis of trigger films or quotes that can be used within the co-design process of future interventions using a experience-based co-design approach.

Participants will also explain how they noticed skin changes in their own skin, to aid in the development of appropriate language and explanations of skin changes in this patient group in an appropriate way.

To achieve the objective each consenting participant will

1. Participate in a semi-structured interview (approx. 1hour) exploring patient experience and patient journey.
2. Self-report their skin tone using Ho and Robinson's skin tones chart, their ethnicity, age & gender.

1.4 Participants 1.4.1 Source of participants.

Participants will be recruited from any of the following :

* through charity organisations such as the "Lyndsey Leg Club Foundation". Publicity for recruitment will be available by adverts circulated through their members lists, on social media or as in person posters at events.
* people who have previously expressed interest in being involved in research on leg ulcers/ venous insufficiency who have a dark skin tone.
* through the "Be Part of Research" network.
* Clinical settings (hospital and community settings).
* Social media adverts 1.4.2 Inclusion / Exclusion Criteria inclusion criteria
* people with chronic venous insufficiency, or their close family member
* the person with chronic venous insufficiency has a dark skin tone (from Ho and Robinson skin tone range 2b-6b).
* ability to give informed consent exclusion criteria
* person with chronic venous insufficiency has a light skin tone (from Ho and Robinson skin tone range 1a-2a, ).
* people unable to speak and understand English
* people unable to give informed consent.

Work package 2 - Informing skin assessment technique and medical photography 2.1 Objective

The primary objective of this work package is to:

• Investigate the efficacy, inter-rater reliability and patient experience of skin assessment techniques in the assessment of skin changes associated with chronic venous disease in people with dark skin tones.

The secondary objective is to:

• determine the acceptability of undergoing these assessments from patient and nurse perspective 2.2 Purpose To explore whether non-invasive assessment (inspection, palpation and skin photography) techniques are appropriate to assess skin changes associated with venous hypertension and chronic venous insufficiency in people with dark skin tones. It will do this by providing proof-of-concept of the use of non-invasive inspection and palpation techniques currently used in practice and techniques recommended by clinical experts. We hope this will improve the evidence base of these techniques. It will also provide proof of concept whether skin photography techniques can be modified to improve skin changes associated with venous hypertension and chronic venous disease on people with dark skin tones. This following suggestions in previous research on skin assessment in people with dark skin tones that modifying the photographs is advantageous to assess for erythema associated with pressure damage in the laboratory setting. However, to date no research has considered whether this could be advantageous to assist in the detection of skin changes associated with CVI, or could be undertaken in the clinical setting.

2.3 Study design This part of the study is an analytical cross-sectional study of 15 patients which includes reviewing participating patients clinical notes. This design enables assessment information to be captured on participating individuals and analyse associations with assessment data from scan results to enable proof-of-concept of skin assessment techniques in people with dark skin tones.

To achieve this objective each consenting participant will

1. undergo the following:

   * a physical assessment of their lower legs using inspection and palpation to determine both their clinical (C) classification of the CEAP and their Venous Clinical Severity Score.
   * answer questions relating to their leg including whether they have noticed any visual skin changes or any changes in symptoms such as pain, itching or sensation
   * wound care photography under standard and enhanced photography techniques in the medical photography studio This data will be compared to their observations taken as part as their clinical care (such as Duplex Scan results, Consultant Diagnosis, ABPI results, CEAP and Venous Clinical Severity Scores reported by the clinical team).
2. Self-report their skin tone using Ho and Robinson's skin tones chart, their ethnicity, age & gender.
3. Give their feedback during a qualitative interview of their experiences of undergoing these clinical assessments based on relevant dimensions of acceptability identified by Sekhon and colleagues (affective attitude, burden, ethicality, perceived effectiveness), and report any adverse events they experienced when undertaking these additional assessments.

The research nurse will also give their feedback of undertaking the assessments on each patient in their structured field notes documenting relevant dimensions of acceptability identified by Sekhon and colleagues (affective attitude, perceived effectiveness, self-efficacy).

2.4 Participants 2.4.1 Source of participants. Participants will be recruited from a clinical setting 2.4.2 Inclusion / Exclusion Criteria inclusion criteria

* people diagnosed with chronic venous insufficiency at NHS trust
* people with a dark skin tones (from Ho and Robinson skin tone range 2b-6b).
* ability to give informed consent
* either coming back to the hospital for surgery or being able to travel back to the hospital to undergo physical assessment and skin photography prior to any intervention.
* have duplex scan results to show blood flow in their leg(s) exclusion criteria
* person with chronic venous insufficiency has a light skin tones (from Ho and Robinson skin tone range 1a-2a).
* people unable to speak and understand English
* people unable to give informed consent.

ELIGIBILITY:
Work-package 1 - Mapping patient journeys and patient experiences Participant inclusion criteria

* people with chronic venous insufficiency, or their close family member
* the person with chronic venous insufficiency has a dark skin tone (from Ho and Robinson skin tone range 2b-6b, table 1).
* ability to give informed consent Participant exclusion criteria
* person with chronic venous insufficiency has a light skin tone (from Ho and Robinson skin tone range 1a-2a, table 1).
* people unable to speak and understand English
* people unable to give informed consent.

Work package 2 - Informing skin assessment technique and medical photography Participant inclusion criteria

* people diagnosed with chronic venous insufficiency at NHS trust
* people with a dark skin tones (from Ho and Robinson skin tone range 2b-6b, table 1).
* ability to give informed consent
* either coming back to the hospital for surgery or being able to travel back to the hospital to undergo physical assessment and skin photography prior to any intervention.
* have duplex ultra-sound scan informing clinical diagnosis of venous disease. Participant exclusion criteria
* person with chronic venous insufficiency has a light skin tones (from Ho and Robinson skin tone range 1a-2a, table 1).
* people unable to speak and understand English
* people unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Work-package 1 - Mapping patient journeys and patient experiences Source of participants.
  People with with chronic venous insufficiency, or their close family member, will be recruited from any of the following :
  * through charity organisations such as the "Lyndsey Leg Club Foundation". Publicity for recruitment will be available by adverts circulated through their members lists, on social media or as in person posters at events.
  * people who have previously expressed interest in being involved in research on leg ulcers/ venous insufficiency who have a dark skin tone.
  * Clinical settings (community or acute setting).
  Work package 2 - Informing skin assessment technique and medical photography Source of participants. Participants will be recruited from clinical settings within our trust partner organization. This NHS Foundation Trust is the hub of the southeast Thames vascular network, based in London, UK.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Work-package 1 - Patient experience | Baseline
  No quantitative outcomes will be assessed in the interview study to map patient journey and patient experience.
Work package 2 - Skin assessment of the lower limb | Baseline
  the clinical researcher / research nurse will follow guidance on assessing the skin in people with dark skin tones. The current guidance on this includes using touch (palpation) as well as visualising skin changes to feel for any temperature change or tightness, and asking the patient whether they have noticed any changes in appearance of have any symptoms such as pain, itching or sensation changes. Al In addition to the assessments recommended in existing clinical guidelines, there is an indication from our recent qualitative interviews with specialist staff, some clinicians have refined their skills and techniques to assist them to undertake, what they perceive to be, a more accurate assessment on people with dark skin tones. This includes several techniques that have not been reported elsewhere including the use of transillumination and extending the skin to visualize changes.
  All these assessments will be reported for each patient.
Work package 2 - Clinical (C) classification of the CEAP | Baseline
  This assessment will be based on the Clinical (C) classification of the CEAP, which is the most widely used tool for venous disease classification and recommended by international guidelines. These may not be readily observed in patients with dark skin tones, especially by non-specialist clinicians. The clinical researcher / research nurse will base their clinical interpretation of CEAP score based on their assessments of skin changes. Individual observations will be reported alongside the classification assigned.
  This scale denotes clinical classification of skin changes from C0 (no visible or palpable signs of venous disease) to C6 (an active venous ulcer).
Work package 2 - Venous Clinical Severity Score | Baseline
  This is a a widely used tool for rating clinical severity which guidance suggests should be considered in research on venous disease. The clinical researcher / research nurse will base their clinical interpretation of each component of the venous clinical severity score based on their assessments of skin changes and patient assessment. Individual observations will be reported alongside the classifications assigned.
  This scale scores several components such as pain, varicose veins, venous oedema, pigmentation, inflammation, induration, active ulcers, use of compression. Each question can score between 0 and 3 points, where more points equates to more severe.
Work package 2 - Wound photography under standard and modified conditions | Baseline
  These images will provide proof of concept whether skin photography techniques can be modified to improve skin changes associated with venous hypertension and chronic venous disease on people with dark skin tones. This following suggestions in previous research on skin assessment in people with dark skin tones that modifying the photographs is advantageous to assess for erythema associated with pressure damage in the laboratory setting. However, to date no research has considered whether this could be advantageous to assist in the detection of skin changes associated with CVI, or could be undertaken in the clinical setting.

SECONDARY OUTCOMES:
Work package 2 - Patient experience | Follow up (less than 72 hours after data obtained)
  Patient perspective of undertaking these assessments. It will explore what they felt of these assessments to ensure patients feel these assessments are appropriate, they felt these are effective and whether they caused any unnecessary discomfort or inconvenience. Data will be collected qualitatively to capture patients perceptions, feelings and opinions.
Work package 2 - Clinican experience | Follow up (less than 24 hours after data obtained)
  Give their feedback of undertaking the assessments on each patient in their structured field notes

CONTACTS AND LOCATIONS:
Overall Officials: Victoria J Clemett, PhD, BNurs, Principal Investigator — King' College London
Locations (2):
- United Kingdom (2):
  - Guy's and St Thomas' NHS Foundation Trust, London, London
  - King's College London, London

IPD SHARING:
Plan to Share IPD: Yes
Data collected as part of this study will be stored in King's Open Research Data System (KORDS), providing long-term storage. This enables DOIs issued for long-term access and citation.
Supporting Information: Study Protocol
Time Frame: The study protocol will be available once ethical approval is granted.